CLINICAL TRIAL: NCT02871453
Title: Scalp Acupuncture for Motor Dysfunction in Ischemic Stroke: a Randomized, Controlled Trial
Brief Title: Evaluating the Therapeutic Effect of Scalp Acupuncture Treatment for Motor Dysfunction in Ischemic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZYSNXD-CC-HPGC-JD-004
Record Dates: First submitted 2016-07-17; First posted 2016-08-18 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Ischemic Stroke; Hemiplegia
Keywords: Ischemic Stroke; Motor Dysfunction; Scalp Acupuncture
MeSH Terms: conditions — Ischemic Stroke; Hemiplegia; Neurologic Manifestations | interventions — Acupuncture Therapy; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture combined rehabilitation (Experimental): Scalp acupuncture treatment
  Rehabilitation treatment
  Interventions: Device: Scalp Acupuncture Treatment
- Rehabilitation (Experimental): Rehabilitation treatment
  Interventions: Other: Rehabilitation treatment

INTERVENTIONS:
Device: Scalp Acupuncture Treatment — The Motor Area of the scalp acupuncture is located over the anterior central convolution of the cerebral cortex, being a line starting from a point 0.5cm posterior to the midpoint of the anterior-posterior midline of the head and stretching diagonally to the juncture between the eyebrow-occipital line and the anterior border of the corner of temporal hairline is indistinct, draw a vertical line upward from the middle point of the zygomatic arch to the eyebrow-occipital line, the intersection of the two lines is the projection of the Motor Area. Needles will be inserted in an about 15 degree angle to a depth of 1.0-1.5cm. Needles are rotated at least 200 revolutions per minute for 1 minute every 10 minutes for a total of 60 minutes. five times a week, 8 weeks in total.
  Other Names: Acupuncture
  Arms: Acupuncture combined rehabilitation
Other: Rehabilitation treatment — The rehabilitation program was designed according to the Chinese stroke rehabilitation treatment guidelines, which included physical therapy (PT) and occupational therapy (OT). The rehabilitation programs will be carried out five times a week (that is, Monday to Friday) for 8 weeks, and every time the rehabilitation treatment( PT and OT) will last approximately for 1 hour. All rehabilitation treatment will be carried out by qualified therapists.
  Arms: Rehabilitation

SUMMARY:
The investigators design a randomized, control study to evaluate the therapeutic effect of scalp acupuncture using Jiao's motor area for motor dysfunction in ischemic stroke patients using the following outcomes: motor function, activity of daily living,quality of life.

DETAILED DESCRIPTION:
Functional disorder is a common and serious consequence of stroke. A large proportion of stroke patients develop motor dysfunction in the early stage after stroke. Acupuncture is often used as an adjunct to mainstream rehabilitation after stroke. Jiao's scalp acupuncture is a contemporary acupuncture technique integrating traditional Chinese needling methods with western medical knowledge of representative areas of the cerebral cortex. It has been widely applied to be a kind of effective treatment for stroke in China. But, there is meta-analysis suggests that with stroke rehabilitation, acupuncture has no additional effect on motor recovery but has a small positive effect on disability, which may be due to a true placebo effect and varied study quality. The efficacy of acupuncture without stroke rehabilitation remains uncertain, mainly because of the poor quality of such studies.

The objective of this proposed study is to determine whether scalp acupuncture treatment could improve significantly motor function in ischemic stroke patients.

In this 8-week, assessor-blind, randomized, controlled study of scalp acupuncture as additional treatment with the rehabilitation treatment, a total of 116 patients with ischemic stroke patients will be recruited. The patients will be randomly assigned to scalp acupuncture combined with rehabilitation treatment (n =58) or rehabilitation treatment (n =58). (40 sessions, 5 sessions a week). Changes in the motor function over time are measured using Fugl-Meyer Scale, Modified Barthel Index and SS-QOL scale. The study will be conducted at Shanghai University of Traditional Chinese Medicine, Long Hua Hospital, Fudan University, Hua Shan Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. The ages of stroke patients from 40 years old to 70 years old
2. Stroke diagnosed according to the criteria of cerebral arterial thrombosis in Western medicine and apoplexy in Chinese medicine
3. Ischemic stroke confirmed by CT brain or MRI brain, with stable medical condition and awareness clear
4. Recent stroke from 1 month to 6 months after onset
5. Stroke with limb motor dysfunction
6. Sufficient cognition to follow commands and Mini-Mental State Examination (MMSE) score > 24
7. Voluntary participation and informed consent signed.

Exclusion Criteria:

1. Stroke with conscious disturbance or serious cognitive impairment
2. Presence of another chronic disorder, including severe Parkinson's disease, cardiac disease, cancers, epilepsy, or chronic alcoholism
3. Impaired hepatic or renal function
4. bleeding tendency
5. Being oversensitive to acupuncture
6. participation in another clinical trial.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline FMA at 4 weeks, 8 weeks | The FMA will be assessed at baseline, interventions period (4 weeks, 8 weeks) and fellow-up period at (1 month, 2 months).
  The Fugl-Meyer Assessment (FMA) scale for motor function, the FMA was developed as the first quantitative evaluative instrument for measuring sensorimotor stroke recovery, which includes an assessment of the upper extremity (UE, 66 points) and lower extremity (LE, 34 points). The motor domain has well-established reliability and validity as an indicator of motor impairment severity across different stroke recovery time points

SECONDARY OUTCOMES:
Change from Baseline MBI at 4 weeks, 8 weeks | The MBI will be assessed at baseline, interventions period (4 weeks, 8 weeks) and fellow-up period at (1 month, 2 months).
  The Barthel Index(BI) is a scale that measures ten basic aspects of activity daily living related to self-care and mobility. For the Chinese Modified Barthel Index(MBI) version, the ten items are: continence of bowels and bladder, feeding, dressing, transferring to and from a toilet, grooming, bathing, moving from wheelchair to bed and return, walking on level surface for 45 meters, and ascend and descend stairs. Standard for Evaluation：Each item (activity) be divided into 5 levels, different level represents a different degree of independence, the lowest level is 1 and the highest level is 5.The more higher level, more independence. The normal score is 100. If a person score is 100, he is able to get along without attendant care.
Change from Baseline SS-QOL at 4 weeks, 8 weeks | The SS-QOL will be assessed at baseline, interventions period (4 weeks, 8 weeks) and fellow-up period at (1 month, 2 months).
  The Stroke-Specific Quality of Life Scale (SS-QOL) is a patient-reported outcome measure intended to provide an assessment of health-related quality of life, specific to patients with stroke. The SS-QOL questionnaire consists of 49 items in the 12 domains of energy, family roles, language, mobility, mood, personality, self-care, social roles, thinking, upper extremity function, vision, and work. Scoring of the SS-QOL is rated on a 5-point Likert scale. Response options are scored as 5 ("no help needed/no trouble at all/strongly disagree"), 4 ("a little help/a little trouble/moderately disagree"), 3 ("some help/some trouble/neither agree nor disagree"), 2 ("a lot of help/a lot of trouble/moderately agree"), and 1 ("total help/could not do it at all/strongly agree"). The domains are scored separately, and a total score is also calculated, with higher scores indicating better function.
Change from Baseline SSTCM at 4 weeks, 8 weeks | The SSTCM will be assessed at baseline, interventions period (4 weeks, 8 weeks) and fellow-up period at (1 month, 2 months).
  The Stroke Syndrome of TCM (SSTCM) was developed mainly based on quantified index of TCM symptoms. The SSTCM includes signs and symptoms which were the most concern of the patients and doctors themselves after stroke. SSTCM mainly consists of two domains: TCM symptoms and pulse conditions and tongue pictures. TCM symptoms area contains 24 items. The assessment standards of each item was divided into four levels and corresponding scores (normal = 0, light = 1, middle=2, heavy = 3) according different degree base on the severity of the symptoms and the impacts on life. Pulse conditions and tongue pictures record contents only, not to score. The total score is calculated from the domain one, with lower scores indicating the lighter degree of the symptom severity and the less impact on life. The SSTCM was evaluated by experienced traditional Chinese medicine doctors who were accepted the unification of assessment training.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Pei, MD, Study Chair — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Pei J, Khiati D, Fu Q, Cui X, Song Y, Yan M, Shi L, Cai Y, Ma Y. Acupuncture treatment on the motor area of the scalp for motor dysfunction in patients with ischemic stroke: study protocol for a randomized controlled trial. Trials. 2017 Jun 20;18(1):287. doi: 10.1186/s13063-017-2000-x. PMID 28633675